CLINICAL TRIAL: NCT03048396
Title: Transplantation of an Uterus for Treatment of an Absolute Uterine Infertility
Brief Title: Acceptance of Uterus Transplantation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FEH_Uterustransplantation
Record Dates: First submitted 2016-12-31; First posted 2017-02-09 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Resolve Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Uterus transplantation (Experimental)
  Interventions: Procedure: Uterus transplantation

INTERVENTIONS:
Procedure: Uterus transplantation

SUMMARY:
Transplantation of an uterus

DETAILED DESCRIPTION:
Uterus transplantation will be performed from live donors to patients with absolute uterine factor infertility. Organ procurement from the donor will be performed by laparotomy. Transplantation will also be performed by laparotomy. Embryo transfer will be done 10-12 months after transplantation. After birth of 1-3 children the uterus will be removed by hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* age below 40 years
* absolute uterine factor infertility
* BMI < 30

Exclusion Criteria:

* systemic disease
* psychiatric disease

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-10; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who are interested in an uterus transplantation | 3 years
Number of patients from these who do have a potential donor | 3 years
Number of patients from these who do have a medical indication for an uterus transplantation | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sara Brucker, MD, Principal Investigator — Research Institute for Women's Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brucker SY, Brannstrom M, Taran FA, Nadalin S, Konigsrainer A, Rall K, Scholler D, Henes M, Bosmuller H, Fend F, Nikolaou K, Notohamiprodjo M, Rosenberger P, Grasshoff C, Heim E, Kramer B, Reisenauer C, Hoopmann M, Kagan KO, Dahm-Kahler P, Kvarnstrom N, Wallwiener D. Selecting living donors for uterus transplantation: lessons learned from two transplantations resulting in menstrual functionality and another attempt, aborted after organ retrieval. Arch Gynecol Obstet. 2018 Mar;297(3):675-684. doi: 10.1007/s00404-017-4626-z. Epub 2017 Dec 21. PMID 29270725